CLINICAL TRIAL: NCT06949176
Title: Clinical Antibacterial Efficacy and Treatment Outcome After Implementing Various Root Canal Irrigating Procedures
Brief Title: Clinical Investigation of Chemomechanical Parameters for an Efficient Disinfection of the Root Canal
Acronym: ENDOA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Giorgos Tzanetakis, Associate Professor, Department of Endodontics, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 594/07.06.2023
Record Dates: First submitted 2025-04-01; First posted 2025-04-29 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Apical Periodontitis; Root Canal Infection
Keywords: apical periodontitis; copious irrigation; mechanical root canal preparation
MeSH Terms: conditions — Periapical Periodontitis | interventions — Sodium Hypochlorite; Hydrogen Peroxide; sodium sulfate

STUDY DESIGN:
Intervention Model Description: The present research will be designed as two-arm, parallel, randomized clinical study. The randomization of the teeth for sampling will be performed through the use of a special software . All the treatment and sampling procedures will be carried out by the same investigator (PhD candidate Dr. Agapi Zervaki).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group A (2,5% NaOCl concentration) (Experimental): Group A will be formed by 22 patients and each teeth will receive 2,5% NaOCl . Working length (WL) will be established according to apex locator (Root ZX mini, Morita). Chemomechanical preparation will be completed in the same appointment.
  Interventions: Procedure: Root canal tratment using mecchanical and chemical preparation.; Drug: Sodium Hypochlorite.; Drug: Hydrogen peroxide.; Drug: Sodium Sulfate.
- Experimental group B (5% NaOCl concentration) (Experimental): Group B will be formed by 22 patients and each teeth will receive 5 % NaOCl .
  Interventions: Device: Root ZX mini apex locator (Morita).; Device: Protaper Gold rotary files (Dentslpy Maillefer).; Device: Smarttrack and Hyflex totary files.; Device: Endo-Eze 27G irrigation needle (Ultradent).

INTERVENTIONS:
Procedure: Root canal tratment using mecchanical and chemical preparation. — Root canal procedures including access cavity preparation, chemomechanical instrumentation, irrigation with sodium hypoclorite (NaOCl), microbiological sampling and obturation with warm vertical compaction.
  Other Names: Endodontic thereapy.
  Arms: Experimental group A (2,5% NaOCl concentration)
Drug: Sodium Hypochlorite. — Sodium Hypoclorite used as the primary irrigant in the root canal treatment at concentrations of 2.5% (Group A) and 5% (Group B).
  Other Names: NaOCl
  Arms: Experimental group A (2,5% NaOCl concentration)
Drug: Hydrogen peroxide. — Applied to the operating field and tooth as part of initial disinfection prior to cavity access.
  Other Names: H202
  Arms: Experimental group A (2,5% NaOCl concentration)
Drug: Sodium Sulfate. — Used to inactivate sodium hypoclorite prior to sample collection.
  Other Names: Na2S2O3
  Arms: Experimental group A (2,5% NaOCl concentration)
Device: Root ZX mini apex locator (Morita). — Used to determine the working length of the root canal.
  Other Names: Morita apex locator.
  Arms: Experimental group B (5% NaOCl concentration)
Device: Protaper Gold rotary files (Dentslpy Maillefer). — Used for coronal flaring in root canal instrumentation.
  Other Names: Dentsply Maillefer rotary system.
  Arms: Experimental group B (5% NaOCl concentration)
Device: Smarttrack and Hyflex totary files. — Used for root canal instrumentation to full working length.
  Other Names: Nikinc and Coltene/Whaledent rotary systems.
  Arms: Experimental group B (5% NaOCl concentration)
Device: Endo-Eze 27G irrigation needle (Ultradent). — Used to deliver irrigant into the root canal.
  Other Names: 27G Luer Lock needle.
  Arms: Experimental group B (5% NaOCl concentration)

SUMMARY:
The aim of the study is first, to evaluate the clinical antibacterial efficacy of two different NaOCl concentrations (2,5% and 5%) under a predefined irrigant flow rate in teeth with pulp necrosis and apical periodontitis by using Real-time PCR. . Second, to evaluate the efficacy of final irrigation by assessing, if possible, a numerical definition for that "so called" as "copious irrigation".

Besides the total microbial load, the antibacterial efficacy of final irrigation procedure against two different bacterial species (namely Pseudoramibacter alactolyticus and Treponema denticola) will also be examined.

DETAILED DESCRIPTION:
The antibacterial efficacy of two different NaOCl concentrations (2,5% and 5%) under a predefined irrigant flow rate in teeth with pulp necrosis and apical periodontitis will be examined through the calculation of the total bacterial load before any treatment procedure and the possible bacteria reduction after each treatment procedure (chemomechanical preparation, and final irrigation treatments). In addition, the antimicrobial efficacy of the above two different concentrations of NaOCl will be compared in terms of treatment outcome. All patients will be asked for one-year recall examination where the outcome of endodontic treatment will be evaluated through clinical and radiographic examination. For the identification of the"copious irrigation" the total amount of final irrigation will be divided in two equal parts of volume/ time (15ml for 5 minutes each). Total bacterial load that will remain after chemomechanical preparation will be compared to the number of bacteria calculated after the first and the second part of irrigation. It will be investigated if final irrigation provides to further microbial reduction and whether prolonged irrigation augments the antibacterial effect.

Besides the total microbial load, the antibacterial efficacy of final irrigation procedure against two different bacterial species (namely Pseudoramibacter alactolyticus and Treponema denticola) will also be examined. First, the prevalence of these specific species will be investigated in primary endodontic infections in Greek-living population. In addition, the effect of chemomechanical preparation and final irrigation procedure on the number of these species will be relatively examined though the reduction curves that will be obtained by qPCR.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the patients who wish to participate in the study.
* Single-rooted teeth with pulp necrosis confirmed by pulp sensibility tests, negative response to both cold and electric pulp testing and radiographic evidence of apical periodontitis.
* Teeth with relatively straight canals, complete root development and no pulp canal obliteration.

Exclusion Criteria:

* Patients who have received antibiotic treatment the last 3 months or need chemoprophylaxis for dental treatment.
* Teeth with previous endodontic treatment.
* Teeth with cracks or incomplete vertical root fracture which disturbs the integrity of the pulp chamber walls.
* Teeth with periodontal pocket more than 4mm.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-06-23 (Estimated)

PRIMARY OUTCOMES:
Reduction of total bacterial load after chemomechanical preparation using 2.5% and 5% NaOCl. | DAY 1: Immediately after chemomechanical preparation.
  Clinical antibacterial efficiency of two different NaOCl concentrations (2.5% and 5%) will be assessed by measuring the total bacteria load reduction using qPCR.
  The unit measure is the Log reduction in total Bacterial DNA copies per sample.
Reduction of total bacterial load after chemomechanical preparation using 2.5% and 5% NaOCl. | DAY 1: Immediately after final irrigation.
  Further reduction of total bacterial load after final irrigation using the same two NaOCl concentrations.
  he unit measure is the Log reduction in total Bacterial DNA copies per sample.
Clinical and radiographic treatment success. | 1 year post tratment.
  Comparison of endodontic treatment outcome between the two NaOCl concentrations groups, assessed by clinical exam and periapical index (PAI).
  Unit measure: Number of teeth scored as healed PAI <2 vs not healed PAI>3.
  Scale Information:
  The Periapical Index (PAI) is a radiographic scoring system ranging from 1 to 5, where:
  1 = Normal periapical structures (best outcome) 5 = Severe periodontitis with exacerbating features (worst outcome) Lower scores indicate better healing.

SECONDARY OUTCOMES:
Additional bacterial load reduction between two sequential 15 ml irrigation periods | Beteen 1 and 6 months after samples collection.
  Evaluation of "copious irrigation" effectiveness by measuring bacterial load after each of two equal 15 ml/5 min final irrigation stages.
  Unit of Measure: Log reduction in total bacterial DNA copies per sample
Prevalence of Pseudoramibacter alactolyticus and Treponema denticola in primary infections | Beteen 1 and 6 months after samples collection.)
  Detection and prevalence rate of two specific bacterial species in untreated teeth with apical periodontitis using qPCR.
  Unit of Measure: Presence/absence and DNA copy number
Reduction in P. alactolyticus and T. denticola load after treatment procedures | Beteen 1 and 6 months after samples collection.
  Quantification of bacterial load changes in P. alactolyticus and T. denticola following chemomechanical preparation and final irrigation.
  Unit of measure: Log reduction in species-specific DNA copy numbers

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos Tzanetakis, Principal Investigator — National and Kapodistian University of Athens
Locations (1):
- National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of the study will be available from the corresponding author upon reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: Data requests will be submitted starting 9 months after article publication and the data will be made accessible up to 24 months. Extensions will be considered.
Access Criteria: Access to trial IPD can be requested by qualified investigators whose proposed research has received IRB approval. Data will be available via a data depository following execution of data use agreement.

REFERENCES:
- [Result] Alves FR, Almeida BM, Neves MA, Rocas IN, Siqueira JF Jr. Time-dependent antibacterial effects of the self-adjusting file used with two sodium hypochlorite concentrations. J Endod. 2011 Oct;37(10):1451-5. doi: 10.1016/j.joen.2011.06.001. Epub 2011 Jul 27. PMID 21924201
- [Result] Antunes HS, Rocas IN, Alves FR, Siqueira JF Jr. Total and Specific Bacterial Levels in the Apical Root Canal System of Teeth with Post-treatment Apical Periodontitis. J Endod. 2015 Jul;41(7):1037-42. doi: 10.1016/j.joen.2015.03.008. Epub 2015 Apr 17. PMID 25892512
- [Result] Barbosa-Ribeiro M, Arruda-Vasconcelos R, Louzada LM, Dos Santos DG, Andreote FD, Gomes BPFA. Microbiological analysis of endodontically treated teeth with apical periodontitis before and after endodontic retreatment. Clin Oral Investig. 2021 Apr;25(4):2017-2027. doi: 10.1007/s00784-020-03510-2. Epub 2020 Aug 28. PMID 32860137
- [Result] Cavrini F, Pirani C, Foschi F, Montebugnoli L, Sambri V, Prati C. Detection of Treponema denticola in root canal systems in primary and secondary endodontic infections. A correlation with clinical symptoms. New Microbiol. 2008 Jan;31(1):67-73. PMID 18437843
- [Result] Gazzaneo I, Vieira GCS, Perez AR, Alves FRF, Goncalves LS, Mdala I, Siqueira JF Jr, Rocas IN. Root Canal Disinfection by Single- and Multiple-instrument Systems: Effects of Sodium Hypochlorite Volume, Concentration, and Retention Time. J Endod. 2019 Jun;45(6):736-741. doi: 10.1016/j.joen.2019.02.017. Epub 2019 Apr 10. PMID 30981431
- [Result] Haapasalo M, Shen Y, Wang Z, Gao Y. Irrigation in endodontics. Br Dent J. 2014 Mar;216(6):299-303. doi: 10.1038/sj.bdj.2014.204. PMID 24651335
- [Result] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698
- [Result] Paiva SS, Siqueira JF Jr, Rocas IN, Carmo FL, Ferreira DC, Curvelo JA, Soares RM, Rosado AS. Supplementing the antimicrobial effects of chemomechanical debridement with either passive ultrasonic irrigation or a final rinse with chlorhexidine: a clinical study. J Endod. 2012 Sep;38(9):1202-6. doi: 10.1016/j.joen.2012.06.023. Epub 2012 Jul 25. PMID 22892736
- [Result] Rocas IN, Siqueira JF Jr. Comparison of the in vivo antimicrobial effectiveness of sodium hypochlorite and chlorhexidine used as root canal irrigants: a molecular microbiology study. J Endod. 2011 Feb;37(2):143-50. doi: 10.1016/j.joen.2010.11.006. PMID 21238793
- [Result] Rocas IN, Siqueira JF Jr. In vivo antimicrobial effects of endodontic treatment procedures as assessed by molecular microbiologic techniques. J Endod. 2011 Mar;37(3):304-10. doi: 10.1016/j.joen.2010.11.003. Epub 2010 Dec 30. PMID 21329812
- [Result] Rocas IN, Siqueira JF Jr. Characterization of microbiota of root canal-treated teeth with posttreatment disease. J Clin Microbiol. 2012 May;50(5):1721-4. doi: 10.1128/JCM.00531-12. Epub 2012 Mar 7. PMID 22403423
- [Result] Rocas IN, Provenzano JC, Neves MA, Siqueira JF Jr. Disinfecting Effects of Rotary Instrumentation with Either 2.5% Sodium Hypochlorite or 2% Chlorhexidine as the Main Irrigant: A Randomized Clinical Study. J Endod. 2016 Jun;42(6):943-7. doi: 10.1016/j.joen.2016.03.019. Epub 2016 Apr 30. PMID 27142579
- [Result] Rodrigues RCV, Zandi H, Kristoffersen AK, Enersen M, Mdala I, Orstavik D, Rocas IN, Siqueira JF Jr. Influence of the Apical Preparation Size and the Irrigant Type on Bacterial Reduction in Root Canal-treated Teeth with Apical Periodontitis. J Endod. 2017 Jul;43(7):1058-1063. doi: 10.1016/j.joen.2017.02.004. Epub 2017 May 5. PMID 28483164
- [Result] Siqueira JF Jr, Rocas IN. Exploiting molecular methods to explore endodontic infections: Part 1--current molecular technologies for microbiological diagnosis. J Endod. 2005 Jun;31(6):411-23. doi: 10.1097/01.don.0000157989.44949.26. PMID 15917679
- [Result] Siqueira JF Jr, Rocas IN. Pseudoramibacter alactolyticus in primary endodontic infections. J Endod. 2003 Nov;29(11):735-8. doi: 10.1097/00004770-200311000-00012. PMID 14651280

DOCUMENTS (3):
  • Study Protocol (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT06949176/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT06949176/SAP_001.pdf
  • Informed Consent Form (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT06949176/ICF_002.pdf